CLINICAL TRIAL: NCT03770208
Title: A Randomized Control Trial of Intravenous Lidocaine for the Management of Traumatic Rib Fractures: a Single Trauma Centre Trial
Brief Title: RIB PAIN (Rib Fractures Treated With Parental Analgesia With Infused LidocaiNe)
Acronym: RIB PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Ian Ball, Chair, Critical Care Western Research and Scholar Program Director; Consultant, Critical Care Medicine; Assistant Professor, Department of Medicine and Department of Epidemiology & Biostatistics, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPIB0247S
Record Dates: First submitted 2018-09-12; First posted 2018-12-10 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Rib Fracture Multiple; Pain, Chest; Pain, Acute; Respiratory Failure; Thoracic Injuries; Trauma Chest
Keywords: Lidocaine Infusions; Thoracic trauma; Analgesic Management; Rib Fractures; Pain
MeSH Terms: conditions — Chest Pain; Acute Pain; Respiratory Insufficiency; Thoracic Injuries; Rib Fractures; Pain | interventions — Lidocaine; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: RCT, single site, double blinded
Who Masked: Participant, Care Provider, Investigator
Masking Description: All parties involved until the end of trial. Pharmacy will be the only unblinded party as they need to prepare the study drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: Standard Care + Placebo (Placebo Comparator): Standard care (acetaminophen, NSAIDs, opioids, gabapentin) as directed by MRP care team plus IV placebo (Lactated Ringers). Lactated Ringers will be delivered as a "initial bolus" and then run as a continuous infusion to mimic the volume (as per Kg) of study drug for 72-96 hours. Standard care will be determined by the care team with no limitations introduced by the research team. Medications utilized and dosing regimes will be recorded after the intervention.
  Interventions: Drug: Control: Standard Care + Placebo
- Intervention: Lidocaine (Experimental): Standard care (acetaminophen, NSAIDs, opioids, gabapentin) as directed by MRP care team plus IV lidocaine. IV lidocaine will be administered as a bolus dose of 2 mg/kg (maximum dose 100 mg) followed by a 2 mg/kg/hr infusion for 72-96 hrs.
  Interventions: Drug: Intervention: Lidocaine

INTERVENTIONS:
Drug: Intervention: Lidocaine — IV Lidocaine bolus plus infusion. Weight based.
  Other Names: Lidocaine Hydrochloride
  Arms: Intervention: Lidocaine
Drug: Control: Standard Care + Placebo — Placebo IV bolus and infusion. Weight based to mimic lidocaine volume.
  Other Names: Lactated Ringers; Ringer's Lactate
  Arms: Control: Standard Care + Placebo

SUMMARY:
Traumatic rib fractures (RF) are a relatively common occurrence in patients of all ages, with a 10% incidence in all trauma patients and are associated with significant morbidity and mortality. Adequate analgesia is paramount for preventing pulmonary complications and can reduce morbidity and mortality. There is longstanding evidence of lidocaine's effectiveness and safety in the post-operative patient and the investigators hypothesize that this modality may prove to be ideal in trauma patients with RF. Therefore, it is imperative that intravenous lidocaine be investigated to ascertain if there is significant benefit for pain reduction in patients who have sustained rib fractures.

A single-centre, double-blind, randomized control trial to evaluate the analgesic efficacy of a 72-96 hour IV lidocaine infusion plus standard analgesics versus placebo infusion plus standard analgesics will be performed on patients (age 18 or older) diagnosed with two or more traumatic rib fractures ,from blunt thoracic trauma, requiring hospital admission at Victoria Hospital.

The primary outcome is mean pain score, as measured on the Visual Analog Scale (VAS) when the patient is at rest and with movement. Secondary outcomes are protocol adherence, patient satisfaction as measured on the VAS, incidence of respiratory failure requiring mechanical ventilation, hospital length of stay, ICU length of stay, mortality, incidence of lidocaine toxicity, treatment regimens (use of additional non-opioid analgesics) and total morphine equivalents used (including breakthrough doses).

This trial will serve to quantify the analgesic efficacy of intravenous lidocaine for patients with traumatic rib fractures. Successful completion of a single centre trial will inform the development of a multi-centre trial powered to demonstrate a reduction in respiratory failure in the trauma population.

DETAILED DESCRIPTION:
This trial will use a randomized double blind design. All patients (age 18 or older) diagnosed with two or more traumatic rib fractures requiring hospital admission at Victoria Hospital will be identified at the time of admission by trauma team members and / or ICU research assistants. Patients unable to understand or follow instructions in English or French, and those unable to complete the Visual Analog Scale (VAS) for pain for any reason, will be excluded.

Any physician member of the inpatient trauma service team, trauma nurse practitioner, or ICU research assistants may approach patients and their families to discuss participation in the trial. Research assistants will be responsible for providing the Letter of Information and Consent Form to families, and storing them once complete. Consented patients will be randomized at admission using the online randomization tool, like REDCAP, by pharmacy. Once randomized, research assistants will contact pharmacy to order "Study Drug", but will remain blinded to study arm

Consented patients will receive either standard care (acetaminophen, NSAIDs, opioids) plus IV placebo or standard care plus IV lidocaine using a fixed strategy with variable blocks and a 1:1 allocation ratio. The pharmacy will be the only party unblinded to randomization and will distribute the "Study Drug" [either IV lidocaine or Lactated Ringer's (a clear colourless solution that is indistinguishable from Lidocaine)] to study participants. All patients will be followed throughout their hospital stay by our research assistants to assess pain and secondary outcomes.

IV lidocaine will be administered as a bolus dose of 2 mg/kg (maximum dose 100 mg) followed by a 2 mg/kg/hr infusion for 72-96 hrs. Lactated Ringer's will be administered at the same overall rate to the control group. Patient pain scores will be accessed at the bedside using the VAS at time 0hrs and every six hours for the duration of study drug infusion.

Daily monitoring of the patient will be performed by the trauma team and bedside nurses. Clinical care will be conducted as usual with the exception of the provision of study drug, the recording of pain Q6 hours, and the assessment of patient satisfaction at the end of the 72-96 hour infusion. All other patient data will be collected from the patient's EMR and bedside chart. In accordance with LHSC hospital Lidocaine policy, all study patients will be on telemetry to monitor for arrhythmias resulting from lidocaine toxicity. As the use of IV lidocaine is already common in the LHSC patient population, all nursing staff are trained to detect signs and symptoms of lidocaine toxicity, and will contact the treatment and research teams if these develop. The study drug infusions will be stopped if any signs of toxicity are seen. The treating team will be unblinded to randomization group in any cases of suspected Lidocaine toxicity.

The primary outcome will be mean pain score calculated from the multiple VAS measures performed during Lidocaine infusions when the patient is at rest and with movement. Secondary outcomes are protocol adherence, patient satisfaction as measured on the VAS, incidence of respiratory failure requiring mechanical ventilation, hospital length of stay, ICU length of stay, mortality, incidence of lidocaine toxicity, treatment regimens (use of additional non-opioid analgesics) and total morphine equivalents used (including breakthrough doses). Secondary outcomes will be recorded by the ICU research assistants on a daily basis during each patient's index stay. Research assistants will help administer the satisfaction survey to patients as soon as possible following completion of the 72-96 hour Lidocaine infusion. The methodology, pain and satisfaction reporting with VAS is very similar to the investigator's previous work.

A sample size of 26 patients is required to find a difference between two independent group means using the following parameters: (1) a 20% reduction in VAS score (20mm), (2) 90% power, (3) probability of a Type I error = 5%, and s stand deviation of 15% (15mm).

An anticipated attrition rate of 20% will be used to ensure enough patients are included for adequate power. Therefore a minimum of 32 patients will be enrolled in the study.

Continuous data will be reported as mean +/- standard deviation or median and interquartile range, depending on the distribution of each data point. Categorical data will be reported as percentages with corresponding 95% confidence intervals. The mean pain score will be compared between treatment groups using Student's T-test. Findings with a Type I error rate < 5% will be considered statistically significant. Analyses of secondary outcomes will be primarily descriptive. Any significance testing of these outcomes will be strictly hypotheses-generating.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, 18 years or older, admitted to Victoria Hospital's Trauma Service with two or more traumatic rib fractures.

Exclusion Criteria:

* Patients under 18 years old
* Patients who sustained complex trauma with multiple other injuries or have decreased LOC or required intubation at admission
* Patients with a known allergy/sensitivity to Lidocaine or other local anesthetic, amide anesthetics or components of the solution
* Patients with a known history of hypersensitivity to methylparaben and/or propylparaben (preservatives used in multidose solutions), or to their metabolite para amino benzoic acid
* Patients who do not speak English with adequate fluency to consent or participate in the VAS survey
* Patients receiving epidural analgesia for another reason
* Patients with pre-existing cardiac arrhythmias including Adam-Stokes syndrome; Wolff- Parkinson-White syndrome; and severe degrees of sinoatrial, atrioventricular, or intraventricular heart block (except in patients with a functioning artificial pacemaker)
* Patients who are known to be pregnant or breast feeding, as identified on Past Medical History, or by initial laboratory investigations performed as a part of standard trauma team assessment
* Patients with known hepatic/renal disease, as identified on Past Medical History, or by initial laboratory investigations performed as a part of standard trauma team assessment
* Patients who refuse inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean Visual Analogue Scale (VAS) Score for Pain | Pain score to be measured before treatment initiation and every 6 hours thereafter until 72-96 hours. Scores will be performed by bedside nursing.
  The primary outcome will be mean pain score calculated from the multiple VAS measures performed during Lidocaine infusions when the patient is at rest and with movement. The VAS for pain is a continuous numerical scale, demonstrated by a horizontal or vertical line, 10 cm long, with verbal descriptors at each end demonstrating the extremes, +/- a central descriptor. It is a scale essentially from 1 to 10, with one being no pain and 10 being the worst pain possible. Subjects mark on the line their approximate pain score by drawing a transecting line. This will be measured with a ruler from the start point on the line and recorded as a data point.

SECONDARY OUTCOMES:
Incidence of Protocol Non-adherence | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Incidence of protocol violations with corresponding 95% confidence intervals. Descriptions of the deviations will be recorded. Types include, number of patients who received lidocaine that were not assigned to that group; number of patients who were assigned lidocaine and never received the study drug; non-weight based dosages of lidocaine; etc.
Patient satisfaction as measured on the Visual Analogue Scale for Satisfaction | Research assistants will help administer the satisfaction survey to patients as soon as possible following completion of the 72-96 hour Lidocaine infusion.
  The VAS for pain is a continuous numerical scale, demonstrated by a horizontal or vertical line, 10 cm long, with verbal descriptors at each end demonstrating the extremes, +/- a central descriptor. It is measured from one, representing not satisfied at all to ten, representing completely satisfied. Subjects mark on the line their approximate pain score by drawing a transecting line. This will be measured with a ruler from the start point on the line and recorded as a data point. Score will be performed on a VAS at the end of the treatment period.
Incidence of respiratory failure requiring mechanical ventilation | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Categorical data will be reported as percentages with corresponding 95% confidence intervals.
Hospital length of stay | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Continuous data will be reported as mean +/- standard deviation or median and interquartile range, depending on the distribution of each data point.
ICU length of stay | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Continuous data will be reported as mean +/- standard deviation or median and interquartile range, depending on the distribution of each data point.
Incidence of Mortality | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period or when the mortality occurs.
  Categorical data will be reported as percentages with corresponding 95% confidence intervals.
Incidence of lidocaine toxicity/adverse events | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Categorical data will be reported as percentages with corresponding 95% confidence intervals. Toxic symptoms will also be recorded.
Treatment regimens (use of additional non-opioid analgesics): Medication type | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Any non-opioid analgesic medications used will be recorded. Incidence of each medications' use will be reported as percentages with corresponding 95% confidence intervals.
Treatment regimens (use of additional non-opioid analgesics): Dosages | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Dosages of any non-opioid analgesic medications used will be recorded.
Treatment regimens (use of additional non-opioid analgesics): Frequency | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Dosing frequency of any non-opioid analgesic medications used will be recorded.
Treatment regimens (use of additional non-opioid analgesics): Delivery Route | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Route of delivery of any non-opioid analgesic medications used will be recorded. Categories include by mouth (PO); subcutaneously (SubQ); Intravenously (IV); and other.
Total morphine equivalents used (including breakthrough doses) | Will be recorded by the ICU research assistants at the end of each patient's 72-96 hour study period.
  Dose will be the cumulative opioid dose over the 72-96 hour period. Conversion to Morphine Equivalents will be calculated. Continuous data will be reported as mean +/- standard deviation or median and interquartile range, depending on the distribution of each data point.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ball, MD, MSc (Epi), FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayberry JC, Trunkey DD. The fractured rib in chest wall trauma. Chest Surg Clin N Am. 1997 May;7(2):239-61. PMID 9156291
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Sirmali M, Turut H, Topcu S, Gulhan E, Yazici U, Kaya S, Tastepe I. A comprehensive analysis of traumatic rib fractures: morbidity, mortality and management. Eur J Cardiothorac Surg. 2003 Jul;24(1):133-8. doi: 10.1016/s1010-7940(03)00256-2. PMID 12853057
- [Background] Simon BJ, Cushman J, Barraco R, Lane V, Luchette FA, Miglietta M, Roccaforte DJ, Spector R; EAST Practice Management Guidelines Work Group. Pain management guidelines for blunt thoracic trauma. J Trauma. 2005 Nov;59(5):1256-67. doi: 10.1097/01.ta.0000178063.77946.f5. No abstract available. PMID 16385313
- [Background] Wu CL, Jani ND, Perkins FM, Barquist E. Thoracic epidural analgesia versus intravenous patient-controlled analgesia for the treatment of rib fracture pain after motor vehicle crash. J Trauma. 1999 Sep;47(3):564-7. doi: 10.1097/00005373-199909000-00025. PMID 10498316
- [Background] Carrier FM, Turgeon AF, Nicole PC, Trepanier CA, Fergusson DA, Thauvette D, Lessard MR. Effect of epidural analgesia in patients with traumatic rib fractures: a systematic review and meta-analysis of randomized controlled trials. Can J Anaesth. 2009 Mar;56(3):230-42. doi: 10.1007/s12630-009-9052-7. Epub 2009 Feb 11. PMID 19247744
- [Background] Linton DM, Potgieter PD. Conservative management of blunt chest trauma. S Afr Med J. 1982 Jun 12;61(24):917-9. PMID 7046093
- [Background] Pattinson KT. Opioids and the control of respiration. Br J Anaesth. 2008 Jun;100(6):747-58. doi: 10.1093/bja/aen094. Epub 2008 May 1. PMID 18456641
- [Background] Ruppen W, Derry S, McQuay H, Moore RA. Incidence of epidural hematoma, infection, and neurologic injury in obstetric patients with epidural analgesia/anesthesia. Anesthesiology. 2006 Aug;105(2):394-9. doi: 10.1097/00000542-200608000-00023. PMID 16871074
- [Background] Allen DJ, Chae-Kim SH, Trousdale DM. Risks and complications of neuraxial anesthesia and the use of anticoagulation in the surgical patient. Proc (Bayl Univ Med Cent). 2002 Oct;15(4):369-73. doi: 10.1080/08998280.2002.11927867. PMID 16333466
- [Background] Karmakar MK, Ho AM. Acute pain management of patients with multiple fractured ribs. J Trauma. 2003 Mar;54(3):615-25. doi: 10.1097/01.TA.0000053197.40145.62. PMID 12634549
- [Background] Bulger EM, Edwards T, Klotz P, Jurkovich GJ. Epidural analgesia improves outcome after multiple rib fractures. Surgery. 2004 Aug;136(2):426-30. doi: 10.1016/j.surg.2004.05.019. PMID 15300210
- [Background] Arendt K, Segal S. Why epidurals do not always work. Rev Obstet Gynecol. 2008 Spring;1(2):49-55. PMID 18769661
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] Daykin H. The efficacy and safety of intravenous lidocaine for analgesia in the older adult: a literature review. Br J Pain. 2017 Feb;11(1):23-31. doi: 10.1177/2049463716676205. Epub 2016 Oct 24. PMID 28386401
- [Background] Nguyen M, Vandenbroucke F, Roy JD, Beaulieu D, Seal RF, Lapointe R, Dagenais M, Roy A, Massicotte L. Evaluation of the addition of bupivacaine to intrathecal morphine and fentanyl for postoperative pain management in laparascopic liver resection. Reg Anesth Pain Med. 2010 May-Jun;35(3):261-6. doi: 10.1097/AAP.0b013e3181de12e4. PMID 20921837
- [Background] Cherny N, Ripamonti C, Pereira J, Davis C, Fallon M, McQuay H, Mercadante S, Pasternak G, Ventafridda V; Expert Working Group of the European Association of Palliative Care Network. Strategies to manage the adverse effects of oral morphine: an evidence-based report. J Clin Oncol. 2001 May 1;19(9):2542-54. doi: 10.1200/JCO.2001.19.9.2542. PMID 11331334
- [Background] Ball IM, Seabrook J, Desai N, Allen L, Anderson S. Dilute proparacaine for the management of acute corneal injuries in the emergency department. CJEM. 2010 Sep;12(5):389-96. doi: 10.1017/s1481803500012537. PMID 20880433